CLINICAL TRIAL: NCT03708107
Title: Short Term Effects in Pressure-pain Threshold of Percutaneous Galvanic Microcurrent Versus Ischemic Compression in the Trapezius Trigger Points
Brief Title: Percutaneous Microelectrolysis (MEP) Versus Ischemic Compression in Miofascial Trigger Points
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Universitario de Ciencias de la Salud Fundación H.A. Barceló (Other)
Responsible Party: Principal Investigator, Oscar Ronzio, Professor - Researcher, Instituto Universitario de Ciencias de la Salud Fundación H.A. Barceló
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MKC18G11; U1111-1222-0977 (Registry Identifier: Universal Trial Number (UTN))
Record Dates: First submitted 2018-10-11; First posted 2018-10-17 (Actual); Last update posted 2019-12-23 (Actual); Status verified 2019-12

CONDITIONS: Myofascial Trigger Point Pain
Keywords: galvanic current; electrolysis; myofascial trigger point; percutaneous microelectrolysis; dry needling; ischemic compression
MeSH Terms: conditions — Myofascial Pain Syndromes | interventions — Acupressure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The researcher who did the algometry was masked. The researcher who did the statistical analysis was masked.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Percutaneous Microelectrolysis (MEP) (Experimental): Principal MTrP will be detected by digital palpation in the upper trapezius. Algometry will be used to determine if the Pain Pressure Threshold (PPT) is equal or less than 3 KgF/cm2. If not, the patient will be not included. A mark will be done in the MTrP.
  MEP® will be applied with a 0,30 x 25 mm acupuncture needle. The needle will be introduced perpendicularly to the MTrP with 100 uA and then increased up to 600 uA. The current will be paused if the patient feels a burning sensation, pain or oppression, waiting up to the patient feels no discomfort. The procedure will be repeated as many times is necessary until the patient do not feel any discomfort for more than 1 minute.
  Algometry will be done immediately finished the intervention, after 10 minutes and at 24 hs.
  Interventions: Device: MEP
- Ischemic compression (Experimental): Principal MTrP will be detected by digital palpation in the upper trapezius. Algometry will be used to determine if the Pain Pressure Threshold (PPT) is equal or less than 3 KgF/cm2. If not, the patient will be not included. A mark will be done in the MTrP with a marker.
  Ischemic compression will be applied perpendicularly to the MTrP, increasing gradually the pression until the patient refers the maximum tolerable pain. This pressure will be applied for 1 minute.
  Algometry will be done immediately finished the intervention, after 10 minutes and at 24 hs.
  Interventions: Other: Ischemic compression

INTERVENTIONS:
Device: MEP — MEP® will be applied with an acupuncture needle (0,30 x 25 mm). The needle will be introduced perpendicularly to the MTrP with 100 uA and then increased up to 600 uA. The current will be paused if the patient feels a burning sensation, pain or oppression, waiting up to the patient feels no discomfort. The procedure will be repeated as many times is necessary until the patient do not feel any discomfort for more than 1 minute.
  Other Names: Percutaneous microelectrolysis; Percutaneous galvanic microcurrent
  Arms: Percutaneous Microelectrolysis (MEP)
Other: Ischemic compression — Ischemic compression will be applied perpendicularly to the MTrP, increasing gradually the pression until the patient refers the maximum tolerable pain. This pressure will be applied for 1 minute.
  Arms: Ischemic compression

SUMMARY:
The Percutaneous Microelectrolysis ® (MEP®) is a technique that employs a galvanic current up to 990 uA, which is applied percutaneously with an acupuncture needle connected to the cathode. Although it is used in tendinopathies, trigger points and muscle injuries, among other conditions, its bases are mostly empirical and there is lack of evidence.

Ischemic compression is a manual therapy that is usually applied in muscle pain.

Myofascial Pain Syndrome (MPS) usually presents painful myofascial trigger points (MTrPs). One methodology used to quantify the pain in MPS is the algometry, which measures the pressure pain threshold (PPT).

The aim of this study was to compare the effects of MEP® with ischemic compression on MTrPs with algometry.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Between 18 to 30 years old.
* Who referred MTrP in the upper trapezious.
* PPT equal or less than 3 KgF/cm2

Exclusion Criteria:

* Being pregnant.
* Taking analgesic medication at least 24 hours before the intervention.
* Being in physical therapy treatment.
* Needle phobia.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-10-22 (Actual); Primary Completion 2019-12-10 (Actual); Study Completion 2019-12-10 (Actual)

PRIMARY OUTCOMES:
Preasure Pain Threshold (PPT) | 24 hours
  Algometry is used to measure the Preasure Pain Threshold (PPT). PPT is defined as the minimum force applied which induces pain. It was applied in the Miofascial Trigger points.

CONTACTS AND LOCATIONS:
Overall Officials: Oscar Ronzio, Study Director — I.U. Fundación H.A. Barceló - U. Maimónides - U. Nacional Arturo Jauretche
Locations (1):
- Oscar Ronzio, Ciudad Autónoma de Buenos Aire, Buenos Aires F.D., Argentina

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at www.mepsport.com
Supporting Information: Study Protocol, ICF
Time Frame: After the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and researchers on IPD and clinical study documents from clinical trials supporting products submitted, for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: http://www.mepsport.com